CLINICAL TRIAL: NCT04645277
Title: Clinical Research on Patients With Hemifacial Spasm by Multi-planar Reconstruction, Curved Planar Reconstruction and Magnetic Resonance Virtual Endoscopy
Brief Title: Magnetic Resonance Imaging Study on Patients With Hemifacial Spasm
Acronym: MRI-HFS
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2020-017
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hemifacial Spasm; Magnetic Resonance Imaging
Keywords: Curved Planar Reconstruction; Magnetic Resonance Virtual Endoscopy
MeSH Terms: conditions — Hemifacial Spasm | interventions — Radionuclide Imaging; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MRI using two dimensional reconstruction
  Interventions: Device: Scanning with magnetic resonance imaging
- Patients with MRI using three dimensional reconstruction
  Interventions: Device: Scanning with magnetic resonance imaging

INTERVENTIONS:
Device: Scanning with magnetic resonance imaging — Facial nerves and adjacent blood vessels are scanned using MRI in the patients with hemifacial spasm (HFS). Then multiplanar reconstruction (two dimensional), along with curved planar reconstruction and magnetic resonance virtual endoscopy (three dimensional), will be performed in the different groups of HFS.

SUMMARY:
Up to now, multiplanar reconstruction (MPR) has been widely used to detect the neurovascular compressions (NVC) on the patients with hemifacial spasm (HFS). However, due to lack of stereoscopic vision, this traditional method sometimes can not meet the requirement on identifying the details of NVC, especially when the aberrant vessels turn out to be veins not arteries. The three dimensional analytic techniques, such as curved planar reconstruction (CPR) and magnetic resonance virtual endoscopy (MRVE), may be helpful to improve the sensitivity and specificity on the demonstration of NVC with stereo and dynamic views, so as to assist the design of the surgical plan.

Furthermore, the frequent finding of NVC on MRI studies of asymptomatic patients incited the creation of several strict criteria for the imaging diagnosis of NVC: the vessel must cross perpendicular to the long axis of the nerve, the nerve must be deviated or indented at the root entry zoon (REZ) by the vessel. Alternatively, morphological measurement of the nerve may correlate with the severity of facial spasm due to atrophy of the nerve in most cases of HFS, and is likely secondary to the micro-structural abnormalities, such as axonal loss, demyelination, collagen deposition, etc. In this study, cross-sectional area (CSA) and volume (V) of the cisternal facial nerve will be assessed to determine whether it can be a useful biomarker for predicting the degree of HFS.

ELIGIBILITY:
Inclusion Criteria:

* Primary HFS patients according to medical history and typical facial muscle spasms that are unilateral, involuntary, and had intermittent contractions innervated by the ipsilateral facial nerve. The patient has 1 year disease duration at least.

Exclusion Criteria:

* Secondary causes of HFS, such as tumors or cysts compressing the facial nerve in the cerebellar pontine cistern; Precarious general health status; Percutaneous lesions or surgical treatments; Cardiac pacemaker or metal implants.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary hemifacial spasm patients, the typical symptoms are unilateral, involuntary, and intermittent contractions of facial muscles innervated by the ipsilateral facial nerve.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Detection of Neurovascular Compression by Multiplanar Reconstruction (MPR) Compared with Surgical Findings | 2021.1-2023.1
  Severity of neurovascular compression, which will be judged by MPR, is defined as follows: 1 = no compression; 2 = contact by a vessel; 3 = indentation by a vessel; and 4 = nerve displacement or distortion by a vessel, and the results of MPR need to be compared with the intraoperative findings to obtain the sensitivity and specificity, respectively.
Sensitivity and Specificity of Detection of Neurovascular Compression by Curved Planar Reconstruction (CPR) Compared with Surgical Findings | 2021.1-2023.1
  Severity of neurovascular compression, which will be judged by CPR, is the same criterion as that in the Outcome 1, and the results of CPR need to be compared with the intraoperative findings to obtain the sensitivity and specificity, respectively.
Sensitivity and Specificity of Detection of Neurovascular Compression by Magnetic Resonance Virtual Endoscopy (MRVE) Compared with Surgical Findings | 2021.1-2023.1
  Severity of neurovascular compression, which will be judged by MRVE, is the same criterion as that in the Outcome 1, and the results of MRVE need to be compared with the intraoperative findings to obtain the sensitivity and specificity, respectively.

SECONDARY OUTCOMES:
Change of Facial Nerve Volume (V) from Baseline to 3 years later | 2021.1-2024.1
  Baseline V (mm3) refers to the volume of the cisternal facial nerve prior to the surgical treatment. Meanwhile, the study endpoint is 3 years after the operation, which need another measurement of V.
  Measurements of V will be performed using Medical Image Processing, Analysis, and Visualization software (MIPAV, http://mipav.cit.nih.gov/). The measurements start from the point where the nerves enter the pons to an imaginary demarcation made at the entrance of the nerves into internal acoustic meatus. The facial nerves are manually delineated in each traverse section. The V will be automatically calculated with the MIPAV software.
Change of Facial Nerve Cross Sectional Area (CSA) from Baseline to 3 years later | 2021.1-2024.1
  Baseline CSA (mm2) refers to the cross sectional area of the cisternal facial nerve prior to the surgical treatment. Meanwhile, the study endpoint is 3 years after the operation, which need another measurement of CSA.
  The CSA is calculated at 5 mm from the entry of the facial nerve into the pons in an image plane perfectly perpendicular to the course of each nerve, which also need using a mouse-driven cursor in MIPAV software.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, M.D. & Ph.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Haller S, Etienne L, Kovari E, Varoquaux AD, Urbach H, Becker M. Imaging of Neurovascular Compression Syndromes: Trigeminal Neuralgia, Hemifacial Spasm, Vestibular Paroxysmia, and Glossopharyngeal Neuralgia. AJNR Am J Neuroradiol. 2016 Aug;37(8):1384-92. doi: 10.3174/ajnr.A4683. Epub 2016 Feb 18. PMID 26892985
- [Result] Zhang P, Selim MH, Wang H, Kuang W, Wu M, Ji C, Hu G, Wu L, Zhu X, Guo H. Intraoperative Measuring of the Offending Vessel's Pressure on the Facial Nerve at Root Exit Zone in Patients with Hemifacial Spasm During Microvascular Decompression: A Prospective Study. World Neurosurg. 2019 Feb;122:e89-e95. doi: 10.1016/j.wneu.2018.09.080. Epub 2018 Sep 25. PMID 30261393
- [Result] Naraghi R, Tanrikulu L, Troescher-Weber R, Bischoff B, Hecht M, Buchfelder M, Hastreiter P. Classification of neurovascular compression in typical hemifacial spasm: three-dimensional visualization of the facial and the vestibulocochlear nerves. J Neurosurg. 2007 Dec;107(6):1154-63. doi: 10.3171/JNS-07/12/1154. PMID 18077953
- [Result] Takao T, Oishi M, Fukuda M, Ishida G, Sato M, Fujii Y. Three-dimensional visualization of neurovascular compression: presurgical use of virtual endoscopy created from magnetic resonance imaging. Neurosurgery. 2008 Jul;63(1 Suppl 1):ONS139-45; discussion ONS145-6. doi: 10.1227/01.neu.0000335028.77779.7c. PMID 18728591